CLINICAL TRIAL: NCT06394518
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single-Dose and Multiple-Dose Continuous Intravenous Infusions of TNP-2092 for Injection in Healthy Chinese Participants
Brief Title: Phase 1, Single-Dose and Multiple-Dose Continuous Intravenous Infusions of TNP-2092 for Injection in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2092-IV-09
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Acute Bacterial Skin and Skin Structure Infection (ABSSSI); Prosthetic Joints Infection (PJI)
MeSH Terms: interventions — TNP-2092; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 200 mg single dose group (low-dose group) (Experimental): Participants in the single-dose groups (200 mg in the low-dose group) were enrolled and received a single intravenous infusion of TNP-2092 for injection(Day 1) over 60 min (± 1 0 min).
  Interventions: Drug: TNP-2092 for injection; Drug: placebo
- 300 mg single and multiple dose continuous dose group (medium-dose group) (Experimental): Participants in the single-dose, multiple-dose continuous dosing group (300 mg in the medium-dose group) received a single intravenous infusion of TNP-2092 for injection on Day 1 of the study. Subsequently, TNP-2092 for injection or placebo was administered as an intravenous infusion every 12 hours (q12 h, ± 10 min) daily on Study Days 4 to 10, and the last dose of TNP-2092 for injection was administered on the morning of Study Day 11.
  Interventions: Drug: TNP-2092 for injection; Drug: placebo
- 400 mg single dose group (high-dose group) (Experimental): Participants in the single-dose groups (400 mg in the high-dose group) were enrolled and received a single intravenous infusion of TNP-2092 for injection over 60 min (± 1 0 min)
  Interventions: Drug: TNP-2092 for injection; Drug: placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TNP-2092 for injection — The study had 3 dose groups, a 200 mg single dose group (low-dose group), a 300 mg single and multiple dose continuous dose group (medium-dose group), and 400 mg single dose group (high-dose group)
  Other Names: Rifaquizinone
  Arms: 200 mg single dose group (low-dose group); 300 mg single and multiple dose continuous dose group (medium-dose group); 400 mg single dose group (high-dose group)
Drug: placebo — The placebo for TNP-2092 active drug

SUMMARY:
This is a phase 1, single-center, randomized, double-blind, placebo-controlled, dose-escalation clinical trial of single and multiple intravenous doses of TNP-2092 for injection in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen to 45 years of age, inclusive, of either gender.
* A body weight of at least 50 kg (male participants) or 45 kg (female participants). A Body Mass Index (BMI) of between 18 to 28 kg/m2, inclusive.
* Physical examinations, vital signs, and clinical laboratory tests are normal, or non-clinically significant abnormal judged by Investigator.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* History or clinical manifestations of significant central nervous system, cardiovascular, pulmonary, hepatic, renal, metabolic, other gastrointestinal, urological, endocrine or hematological disease that, in the opinion of the investigator, would confound the study results or compromise subject safety.
* History or presence of alcohol or drug abuse, or illegal drug use.
* Loss or donation of blood (> 450 mL) within 3 months prior to the start of the Screening Period.
* Any history of allergic drug reactions, or any contraindication to the use of rifampin/rifamycin or a fluoroquinolone.
* Taking any medication known to induce or inhibit CYP enzymes within 28 days prior to screening.
* Taking any prescribed or over-the-counter medications within 2 weeks prior to screening, or during the trial, including vitamins, food supplements, herbal remedies, or traditional Chinese remedies.
* Significant abnormal findings on clinical laboratory tests, in the opinion of the Investigator, could jeopardize achieving the study objectives and/or compromise the participant's safety, including but not limited to:

  1. Hematology: hemoglobin (HGB), white blood cell (WBC), absolute neutrophil count (ANC), or platelet count (PLT) < the lower limit of normal (LLN).
  2. Liver function: aspartate aminotransferase (AST) > the upper limit of normal (ULN), and/or alanine aminotransferase (ALT) > ULN, and/or total bilirubin > ULN.
  3. Renal function: serum creatinine > ULN.
* Tests positive for the human immunodeficiency virus (HIV) antibody, treponema pallidum antibody, hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody, and/or urine drug screening.
* Abnormal findings on vital signs, in the opinion of the Investigator, could jeopardize achieving the study objectives and/or compromise the participant's safety, including but not limited to:

  1. Body temperature (ear) ≥ 37.5 ºC.
  2. Blood pressure >140/90 mmHg, or <90/60 mmHg.
  3. Pulse rate > 100 beat/min, or < 50 beat/min.
* Abnormal findings on CT scan of chest and abdominal ultrasonography, in the opinion of the Investigator, could jeopardize achieving the study objectives and/or compromise the participant's safety.
* Any ECG abnormality considered to be clinically significant by the Investigator, or QTcF interval (QT interval corrected for heart rate per Fridericia's formula) > 450 msec.
* Abnormal findings on physical examination, in the opinion of the Investigator, could jeopardize achieving the study objectives and/or compromise the participant's safety.
* Smoking, or consuming coffee, tea, cola, chocolate, grapefruit/grapefruit juice, or alcohol within 48 hours prior to the first dose of the study drug.
* Use of ≥ 5 cigarettes per day within 3 months prior to screening. Participants may not smoking during the study.
* Consume ≥ 14 units of alcohol (1 unit = 285 mL beer, or 25 mL hard liquor/spirits, or 100 mL wine) per week within 6 months prior to screening; or cannot stop consumption of alcohol during the study.
* Received any investigational medication or participated any clinical study within 3 months prior to signing ICF.
* If female, the participant is pregnant, lactating, or serum pregnancy test positive during the screening.
* Cannot abstinence or effective methods of birth control, including his/her partner, during the study and within 12 weeks after the last dose of study drug.
* Venous access considered inadequate for PK sample collection; history or evidence of adverse symptoms associated with phlebotomy or blood donation.
* Any other reason that, in the opinion of the Investigator, would render the subject unsuitable for study enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Day 1 to Day 14
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) | 10, 20, 30, 45 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72 hours after the end of infusion
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma pharmacokinetic(PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Area Under the Plasma Concentration Versus Time Curve from 0 to the Last Measurable Concentration (AUC0-last) | 10, 20, 30, 45 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72 hours after the end of infusion
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Maximum Observed Plasma Concentration (Cmax) of TNP-2092 | 10, 20, 30, 45 minutes, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72 hours after the end of infusion
  Plasma concentrations of TNP-2092 were measured by a specific and validated assay at specified time points

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No